CLINICAL TRIAL: NCT01099215
Title: An Open-Label Dose Escalation Safety Study of PVS-10200 for the Treatment of Restenosis in Patients Undergoing Minimally Invasive Peripheral Revascularization (TRIUMPH)
Brief Title: Study of PVS-10200 for the Treatment of Restenosis in Patients With Peripheral Artery Disease (TRIUMPH)
Acronym: TRIUMPH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVS 03-001; 2009-011998-32 (EudraCT Number)
Record Dates: First submitted 2010-04-01; First posted 2010-04-06 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; percutaneous transluminal angioplasty; stent; balloon/stent; superficial femoral artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PVS-10200 (Other): Each subject will receive one treatment of PVS-10200 delivered by ultrasound guided injection perivascular to the region of the target lesion within 24 hours of the completed angioplasty and stent placement.
  Interventions: Biological: PVS-10200

INTERVENTIONS:
Biological: PVS-10200 — PVS-10200 is composed of allogeneic human aortic endothelial cells cultured in a gelatin matrix.

SUMMARY:
The purpose of this study is to evaluate the safety of two doses of PVS-10200, an allogeneic cellular therapy, delivered as a single injection following percutaneous transluminal ("balloon") angioplasty and stent placement for the treatment of peripheral artery disease (PAD).

DETAILED DESCRIPTION:
This is an open-label dose escalation safety study of PVS-10200 in 30 subjects with peripheral artery disease (PAD) requiring balloon angioplasty and stent placement in the superficial femoral artery (SFA). The study will be completed sequentially in two dose cohorts of 10 subjects (low dose group, Cohort A) and 20 subjects (high dose group, Cohort B). A Data Safety Monitoring Board (DSMB) will conduct regular safety reviews.

Each subject will receive one treatment of PVS-10200 delivered by ultrasound guided injection to the perivascular region (external to the vessel) of the stented target lesion. The treatment will be administered within 24 hours after balloon angioplasty/stent placement.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed the informed consent document and patient information leaflet.
2. Male and female subject ≥ 18 years of age at the time of consent.
3. If female, the subject is (a) at least 1 year post-menopausal, or (b) surgically sterile, or (c) of child-bearing potential, with a negative serum pregnancy test result prior to study enrollment, who agrees to use adequate contraception for 6 months. Adequate contraception is defined as abstinence or a reliable method of birth control (e.g., a hormonal contraceptive, intra-uterine device, implantable or injectable contraceptives (Norplant® or Depo-Provera®), diaphragm, or condom with spermicide).
4. Subject has symptomatic peripheral arterial disease involving the superficial femoral artery, defined as Fontaine Class IIb, III and IV.
5. Meets anatomic requirements based on biplane digital subtraction angiography performed at the time of intervention including:

   * Stenosis of ≥ 50% or occlusion of the superficial femoral artery, and
   * Target lesion length of ≤ 150 mm, and
   * At least one patent (< 50 % stenosis) tibioperoneal runoff vessel
6. Target lesion is 7-15 cm in length.
7. Subject is expected to stay in the same geographic area for at least 48 weeks.
8. In the opinion of the investigator, the subject is able to understand and is willing to complete the study requirements.
9. Subject is receiving a therapeutic dose of statin therapy (starting minimum of 7 days prior to intervention) and continuing for a minimum of 4 weeks post-intervention.

Exclusion Criteria:

1. Subject has acute limb ischemia.
2. Subject has had prior revascularization of the target lesion.
3. Subject has untreated inflow disease of the ipsilateral pelvic arteries (> 50% stenosis or occlusion).
4. The target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion(s).
5. Subject has an unresolved thrombus within the target vessel.
6. Additional percutaneous interventional procedures (cardiac/peripheral) are planned ≤ 30 days following the study procedure.
7. Subject has suffered a hemorrhagic stroke ≤ 6 mo prior to the study procedure.
8. Subject has a history of bleeding diatheses or coagulopathy.
9. Subject is diagnosed with septicemia at the time of the study procedure.
10. Subject is known to be seropositive for HIV.
11. Subject has some other medical illness that may cause the subject to be non-compliant with the protocol.
12. Subject has a known allergy to bovine or porcine products (i.e., heparin).
13. Subject has a known allergy to collagen/gelatin products.
14. Subject has had a severe reaction to contrast media.
15. Subject has a known allergy or intolerance to anti-platelet medication (e.g., acetylsalicylic acid or clopidogrel) or statin therapy.
16. Subject has a history of IV drug use within 6 months prior to screening.
17. Subject has a documented diagnosis of cancer within 2 years (24 months) prior to screening.
18. Subject is a female who is pregnant, breast-feeding, or plans to become pregnant during the study.
19. Subject is currently participating in another investigational drug, biologic or device trial, plans to participate in another investigational drug, biologic or device study during participation in this study, or has completed participation in another investigational drug, biologic or device trial within the last 30 days. Note: Subjects involved in extended follow-up trials for products that are currently commercially available and used as approved are not considered to be participating investigational trials.
20. Subject is a staff member of any of the participating institutions or relative of a staff member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat, Paris

REFERENCES:
- [Derived] Sevestre MA, Larghero J, Castier Y, Nugent HM, Visonneau S, Alsac JM. Pilot safety study of perivascular injection of tissue-engineered allogeneic aortic endothelial cells in patients undergoing minimally invasive peripheral revascularization. J Vasc Surg. 2014 Jun;59(6):1597-606. doi: 10.1016/j.jvs.2014.01.014. Epub 2014 Mar 7. PMID 24613691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was from 30 March 2010 (first patient's screening visit) to 19 June 2012 (last patient's Week 48 visit). A total of 30 subjects were screened for study eligibility, of whom a total of 21 subjects were registered (i.e., enrolled) and treated with PVS-10200. The study was conducted at 3 study centers in France
Groups:
- Low Dose PVS-10200 (Cohort A): Low dose PVS-10200 (6×10^5 cells/cm lesion)
- High Dose PVS-10200 (Cohort B): High dose PVS-10200 (15×10^5 cells/cm lesion)
Period: Overall Study
Arm/Group | Low Dose PVS-10200 (Cohort A) | High Dose PVS-10200 (Cohort B)
Started | 11 | 10
Completed | 10 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: Low dose PVS-10200 (6×10^5 cells/cm lesion)
- Cohort B: High dose PVS-10200 (15×10^5 cells/cm lesion)
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening
  Years | 61.6 (10.11) | 70.7 (7.67) | 66.0 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 6 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  France | 11 | 10 | 21
Resting Ankle Brachial Index, Leg with Target Lesion [Mean (Standard Deviation); unit: ratio] | 0.954 (0.164) | 0.851 (0.258) | 0.902 (0.217)
Fontaine Classification [Count of Participants; unit: Participants]
  STAGE IIB-MODERATE TO SEVERE CLAUDICATION(<200M) | 10 | 6 | 16
  STAGE IV - ULCERATION OR GANGRENE | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Major Adverse Events (MAEs)
Description: Major Adverse Events are: - Death - Major amputation - Procedural related serious adverse events - Investigational product related serious adverse events
Time Frame: within 4 weeks after study procedure
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants | 0 | 0

2. Secondary Outcome: Incidence of Major Adverse Events (MAEs)
Description: as for outcome 1
Time Frame: within 24 and 48 weeks from study procedure
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  Week 24 | 0 | 0
  Week 48 | 0 | 1

3. Secondary Outcome: Incidence of Serious Adverse Events
Time Frame: Up to 48 weeks from study procedure
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants | 7 | 7

4. Secondary Outcome: Incidence of Adverse Events, Laboratory Abnormalities
Time Frame: Up to 48 weeks from study procedure
Population: Safety Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  Treatment Emergent Adverse Events | 11 | 10
  Clinically Significant Laboratory | 1 | 5

5. Secondary Outcome: Maintenance of Primary Patency of Superficial Femoral Artery (SFA)
Description: Primary patency was defined as duplex ultrasound peak systolic velocity [PSV] ratio ≤2.4.Ultrasound data was obtained for each patient at each time point and had to be considered diagnostic and evaluable by the core lab; if it was not, then this analysis could not be done for that particular subject.
Time Frame: within 4 weeks from study procedure
Population: Intention-to-Treat Population Analysis (Data was not available for all 21 subjects because it includes only ultrasound data obtained that was considered diagnostic and evaluable by the core lab)
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 0 | 0
  YES | 9 | 9

6. Secondary Outcome: Maintenance of Primary Patency of Superficial Femoral Artery (SFA)
Description: as for outcome 5
Time Frame: within 24 weeks from study procedure
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 4 | 4
  YES | 5 | 4

7. Secondary Outcome: Maintenance of Primary Patency of Superficial Femoral Artery (SFA)
Description: as for outcome 5
Time Frame: within 48 weeks from study procedure
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 3 | 3
  YES | 4 | 3

8. Secondary Outcome: Rate of Binary In-stent Restenosis
Description: Binary restenosis relied on duplex ultrasound data with a Yes/No assessment with 0-49% being No (peak systolic velocity [PSV] ratio ≤2.4) and Yes being 50-99% (PSV ratio >2.4), with the PSV ratio calculated as PSV from stenosis divided by the PSV from a normal segment of artery proximal to the stenosis. Ultrasound data was obtained for each patient at each time point and had to be considered diagnostic and evaluable by the core lab; if it was not, then this analysis could not be done for that particular subject.
Time Frame: within 4 weeks from study procedure
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 9 | 9
  YES | 0 | 0

9. Secondary Outcome: Rate of Binary In-stent Restenosis
Description: as for outcome 8
Time Frame: within 24 weeks from study procedure
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 9 | 8
  YES | 0 | 0

10. Secondary Outcome: Rate of Binary In-stent Restenosis
Description: as for outcome 8
Time Frame: within 48 weeks from study procedure
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  NO | 8 | 7
  YES | 0 | 0

11. Secondary Outcome: Number of Patients Requiring Reintervention of Target Lesion / Target Vessel
Description: Survival analysis - outcome reported as patients requiring reintervention of the target lesion / vessel
Time Frame: up to 48 Weeks from study procedure
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants | 4 (15.4%) [29.00 to NA] | 2 (12.6%) [52.86 to 65.43]

12. Secondary Outcome: Resting Ankle-brachial Index
Description: ABI was calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressures in the arm. This test is used to predict the severity of PAD.
Time Frame: within 4, 24 and 48 weeks from study procedure
Population: Intention-to-Treat Population Analysis
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
ratio
  Week 4 | 0.984 (0.128) | 0.887 (0.237)
  Week 24 | 0.948 (0.172) | 0.842 (0.204)
  Week 48 | 0.931 (0.193) | 0.857 (0.226)

13. Secondary Outcome: Changes in Physical Exam
Description: Changes in physical examination were compared to baseline: numbers of subjects presenting any new finding or worsening of abnormal findings compared to the screening examination are reported
Time Frame: within 4, 24 and 48 weeks from baseline
Population: Safety Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  Week 4 | 0 | 3
  Week 24 | 5 | 1
  Week 48 | 3 | 3

14. Secondary Outcome: The Fontaine Class of Peripheral Artery Disease
Description: CLASSIFICATION OF PERIPHERAL ATERIAL DISEASE ACCORDING TO FONTAINE Stage Clinical description I Asymptomatic IIA Mild claudication IIB Moderate -severe claudication III Ischemic rest pain IV Ulceration or gangrene
Time Frame: change from baseline to 4 weeks
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  STAGE IIB (Baseline) to STAGE I (Week 4) | 9 | 5
  STAGE IIB (Baseline) to STAGE IIA (Week 4) | 1 | 1
  STAGE IV (Baseline) to STAGE I (Week 4) | 1 | 0
  STAGE IV (Baseline) to STAGE IV (Week 4) | 0 | 4

15. Secondary Outcome: The Fontaine Class of Peripheral Artery Disease
Description: as for outcome 14
Time Frame: change from baseline to 24 weeks
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  STAGE IIB (Baseline) to STAGE I (Week 24) | 4 | 3
  STAGE IIB (Baseline) to STAGE IIA (Week 24) | 4 | 1
  STAGE IIB (Baseline) to STAGE IIB (Week 24) | 2 | 1
  STAGE IV (Baseline) to STAGE I (Week 24) | 0 | 1
  STAGE IV (Baseline) to STAGE IV (Week 24) | 0 | 2
  Missing | 1 | 2

16. Secondary Outcome: The Fontaine Class of Peripheral Artery Disease
Description: as for outcome 14
Time Frame: change from baseline to 48 weeks
Population: Intention-to-Treat Population Analysis
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 10
participants
  STAGE IIB (Baseline) to STAGE I (Week 48) | 6 | 4
  STAGE IIB (Baseline) to STAGE IIA (Week 48) | 1 | 1
  STAGE IIB (Baseline) to STAGE IIB (Week 48) | 3 | 1
  STAGE IV (Baseline) to STAGE I (Week 48) | 0 | 1
  STAGE IV (Baseline) to STAGE IIB (Week 48) | 0 | 1
  STAGE IV (Baseline) to STAGE IV (Week 48) | 0 | 1
  Missing | 1 | 1

ADVERSE EVENTS:
Time Frame: 30 March 2010 (first patient's screening visit) to 19 June 2012 (last patient's Week 48 visit)
Description: No increase in humoral sensitization seen after PVS-10200 treatment. Positive panel-reactive antibodies (PRA) findings seen at Wk 48 only in 2 subjects who also had positive PRA findings at Screening (i.e., sensitized prior to PVS 10-200 exposure). No treatment-emergent Adverse Events associated with humoral sensitization seen in either subject.
Arm/Group | Cohort A | Cohort B
Serious Adverse Events (participants affected / at risk) | 7/11 | 7/10
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) | Cohort B (N=10)
ANGIOPLASTY (Surgical and medical procedures) | 1 | 0
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 2 | 0
ARTERIAL STENOSIS (Vascular disorders) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 3 | 3
INTERMITTENT CLAUDICATION (Vascular disorders) | 6 | 2
LEG AMPUTATION (Surgical and medical procedures) | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 1
TOE AMPUTATION (Surgical and medical procedures) | 0 | 2
WOUND NECROSIS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) | Cohort B (N=10)
Arterial Restenosis (Injury, poisoning and procedural complications) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 4 | 0
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 3 | 3
Injection Site Haemorrhage (General disorders) | 2 | 0
Intermittent Claudication (Vascular disorders) | 6 | 2
Toe Amputation (Surgical and medical procedures) | 0 | 2

LIMITATIONS AND CAVEATS:
Small patient number, no control arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Company-specific confidentiality agreement